CLINICAL TRIAL: NCT05048641
Title: Effectiveness of Mobile Messenger-initiated Reminder on Biannual Mammography Adherence in Breast Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2021.240
Record Dates: First submitted 2021-08-30; First posted 2021-09-17 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp Reminder group (Experimental): Subjects who are allocated to the intervention group received reminder via WhatsApp Messenger at one month before the scheduled calendar month of biannual mammography follow-up.
  Interventions: Other: Whatsapp reminder
- No Reminder (NR) group (No Intervention): Subjects who are allocated to the NR group received standard-of-care service which is no reminder text messages via WhatsApp Messenger prior to their scheduled repeat mammography and no follow up phone reminder until the completion of the outcome measurement period.

INTERVENTIONS:
Other: Whatsapp reminder — Subjects who are allocated to the intervention group received reminder via WhatsApp Messenger at one month before the scheduled calendar month of biannual mammography follow-up.
  Arms: WhatsApp Reminder group

SUMMARY:
Female breast cancer is the most common cancer and fifth leading cause of cancer death worldwide. In the past decade, breast cancer consistently to be the most common cancer for women in Hong Kong, so much that it accounts for 27% of all female cancers, with 4,600 new cases of breast cancer registration every year and the lifetime breast cancer risk for females is 1 in every 14. At the same time, breast cancer ranks the third in cancer death in Hong Kong, with a five-year relative survival rate of 84%. Regular mammography screening has been shown to reduce the mortality of breast cancer. International guidelines recommend annual or biannual mammography screening for women aged 50 or above.

The adherence to regular mammography screening remains a challenge. Studies had shown that the adherence decreased over time. Mailed and telephone reminder were being proven to be effective tools to increase the adherence to regular breast screening using mammography. However, both mailing and telephone strategies are associated with labor intensity and high cost.

Over the past two decades, the advent of internet and smartphone provided a fertile platform for the development of mobile-health technologies. WhatsApp Messenger is one of the most frequently used free-of-charge mobile messenger that permits users to send secure messages across different device platforms. A recent randomized controlled trial from our team has suggested its clinical utility in improving adherence to regular colorectal cancer screening using fecal immunochemical test. This encouraging data prompted us to investigate the potential role of WhatsApp Messenger in breast cancer screening. We hypothesized that text reminder sent via WhatsApp Messenger improves the longitudinal adherence to biannual mammography in a community-based, opportunistic breast screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women with negative mammography results which are defined as BI-RADS (Breast Imaging-Reporting and Data System) 1 or 2 in the first round of mammography screening of the existing opportunistic breast cancer screening cohort
* Due for second round of biannual follow up of mammography
* Consented to be contacted via WhatsApp Messenger

Exclusion Criteria:

* Those without access to WhatsApp Messenger or disagreed to be contacted via WhatsApp Messenger

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Attendance of the second round of mammography follow up and repeat mammography arrangement. | Through study completion, an average of 2 years
  Primary outcome is the adherence to biannual mammography screening, defined as attendance to the second round of mammography follow up and attendance to the repeat mammography arrangement.

SECONDARY OUTCOMES:
Risk factors of nonadherence based on all available variables of patients' characteristics | Through study completion, an average of 2 years
  Secondary outcomes are the risk factors of nonadherence which will be determined by binary logistic regression analysis using all available variables of patients' characteristics

IPD SHARING:
Plan to Share IPD: No